CLINICAL TRIAL: NCT01943747
Title: Surviving Sepsis Campaign. International Multicentre Prevalence Study on Sepsis.
Brief Title: International Multicentre Prevalence Study on Sepsis
Acronym: IMPRESS
Status: Completed | Type: Observational
Sponsor: European Society of Intensive Care Medicine (Other)
Collaborators: Society of Critical Care Medicine (SCCM) (Unknown)
Responsible Party: Sponsor
Other Study IDs: IMPRESS
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: sepsis; severe sepsis; septic shock; infection; organ dysfunction; quality improvement
MeSH Terms: conditions — Sepsis; Shock, Septic; Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To mark 10 years of the Surviving Sepsis Campaign (SSC), and timed to coincide with World Sepsis Day, on September 13, 2013, the SSC, ESICM and SCCM will be conducting an international point prevalence study of severe sepsis and septic shock. The goal of this project is to determine the world wide burden of severe sepsis and define current practices of sepsis care internationally. The study is a simple data collection exercise for patients presenting with either severe sepsis or septic shock on World Sepsis Day.

DETAILED DESCRIPTION:
De---identified patient---level data will be collected on patients presenting to a participating intensive care unit or emergency department with severe sepsis or septic shock over a 24 hour period from 00:00 to 24:00 November 07, 2013. De---identified data that is already collected as part of routine clinical care will be collected for this study. Data to be collected includes hospital and ICU characteristics, patient characteristics, severity of illness, and adherence to SSC bundle elements and mortality. It will take between 30---60 minutes to collect and enter data for each patient admitted with severe sepsis or septic shock over the 24 hours study period.

ELIGIBILITY:
Inclusion Criteria:

To be eligible patients must have all of the following:

* Must be admitted or transferred to either the ED or an Intensive Care Unit.
* Have a high clinical suspicion of an infection
* Have sepsis as defined by an infection together with two or more SIRS criteria
* Evidence of acute organ dysfunction and/or Shock.

Exclusion Criteria:

* Patients less than 18 years of age
* Patients in whom the sepsis has been present from before the beginning of the study period
* Any patients previously included in the study during the same study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients presenting with either severe sepsis or septic shock
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-11; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
28-Day Mortality | one week

SECONDARY OUTCOMES:
Organ Failure | one week

OTHER OUTCOMES:
Length of Stay in the Hospital | one week

CONTACTS AND LOCATIONS:
Overall Officials: Andrew RHODES, MD, PhD, Principal Investigator — European Society of Intensive Care Medicine
Locations (1):
- All centres willing to contribute are welcome., Brussels, Belgium